CLINICAL TRIAL: NCT04007952
Title: Two-Armed Double-Blinded Registry-Based Randomized Control Trial Comparing Anterior Gastropexy to No Anterior Gastropexy for Paraesophageal Hernia Repair
Brief Title: Anterior Gastropexy vs. No Anterior Gastropexy for Paraesophageal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clayton Petro (Other)
Responsible Party: Sponsor-Investigator, Clayton Petro, Assistant Professor, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-616
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Paraesophageal Hernia; Hiatal Hernia Large
Keywords: paraesophageal hernia; gastropexy; minimally invasive surgery
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Intervention Model Description: This will be a double-blinded, registry-based, randomized control trial comparing anterior gastropexy to no anterior gastropexy in paraesophageal hernia repair. This will be a two-arm trial with intervention 1: intervention 2 and control allocation ratio of 1:1.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be informed regarding the treatment that they received until they complete 1-year follow-up. Imaging will be reviewed at the end of the study period by surgeons who are blinded to treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention 1 (Control) (No Intervention): No anterior gastropexy will be performed.
- Intervention 2 (Treatment) (Experimental): Anterior gastropexy will be performed.
  Interventions: Procedure: Anterior Gastropexy

INTERVENTIONS:
Procedure: Anterior Gastropexy — Two permanent sutures will be introduced into the abdomen and placed along the lesser curvature of the stomach. A suture passer will be used to grasp the ends of the sutures to externalize them at separate fascial punctures. At time of abdominal desufflation, the sutures will be tied and the incision closed per individual surgeon practice.
  Arms: Intervention 2 (Treatment)

SUMMARY:
This study evaluates the effect of anterior gastropexy (one or more sutures fixing the stomach to the inner abdominal wall) on improving durability of paraesophageal hernia repair. Half of participants will receive anterior gastropexy, while the other half will not. The hypothesis is that anterior gastropexy will help to prevent paraesophageal hernias from recurring.

DETAILED DESCRIPTION:
Paraesophageal hernias are hernias in which the stomach and/or other abdominal organs herniate through the diaphragm into the chest. This abnormal anatomy can lead to acid reflux, trouble swallowing, and shortness of breath, and can also be a risk factor for surgical emergencies involving the stomach. For these reasons, the Society of American Gastrointestinal and Endoscopic Surgeons has strongly recommended that all symptomatic paraesophageal hernias be repaired.

These repairs are technically challenging, and the best available evidence suggests that more than half of patients undergoing repair will have radiographic hernia recurrence at 5 years after surgery. There has been suggestion that use of anterior gastropexy - in which suture is used to affix the stomach to the anterior abdomen - may reduce recurrence rates. However, it is uncertain whether this data is reliable. While some surgeons use anterior gastropexy routinely because they believe it reduces recurrence, other surgeons do not use anterior gastropexy due to the concern that patients will have short-term pain at the suture site. This study aims to evaluate the effect of using anterior gastropexy on recurrence rates after paraesophageal hernia repair, compared to not using anterior gastropexy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Able to participate in follow-up
* Symptomatic paraesophageal hernia
* Paraesophageal hernia is at least 5 centimeters in height on upper GI study or endoscopy
* Elective laparoscopic paraesophageal hernia repair (must begin laparoscopic, but may convert to open surgery if needed)
* Crura must be reapproximated at time of surgery

Exclusion Criteria:

* Previous operations of the esophagus or stomach
* Emergent operation for acute gastric volvulus
* Paraesophageal hernia repair with concurrent bariatric procedure or procedure to reduce stomach volume
* Placement of gastrostomy tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Paraesophageal Hernia Recurrence | 1 year
  Either radiographic evidence of hernia recurrence on an upper GI study or need for reoperation secondary to paraesophageal hernia recurrence

SECONDARY OUTCOMES:
Mean Change from Baseline in GERD-HRQL Scores at 30 days and 1 year | 30 day follow up (15-45 days postop) and 1 year follow-up (6-18 months)
  The Gastroesophageal Reflux Disease Health-Related Quality of Life (GERD-HRQL) is a 10-item instrument to quantify symptom severity in gastroesophageal reflux disease. Scores on individual items are summed and may range from 0 to 50, with higher scores indicating greater severity of symptoms and worse quality of life. Additionally, there is a question about global satisfaction with quality of life, which may be answered as "satisfied," "neutral," or "dissatisfied." The percentages of these categories will be reported.
Mean Change from Baseline in Symptom Severity Measured by Visual Analog Scale at 30 days and 1 year | 30 day follow up (15-45 days postop) and 1 year follow-up (6-18 months)
  Eight symptoms that are potentially related to the presence of a paraesophageal hernia will be assessed on a scale ranging from 0 to 10, with higher scores indicating more significant impact on quality of life. Symptoms include regurgitation, chest pain, abdominal pain, nausea, vomiting, postprandial pain, cardiovascular, and pulmonary symptoms. Each symptom will be reported separately.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ponsky J, Rosen M, Fanning A, Malm J. Anterior gastropexy may reduce the recurrence rate after laparoscopic paraesophageal hernia repair. Surg Endosc. 2003 Jul;17(7):1036-41. doi: 10.1007/s00464-002-8765-2. Epub 2003 Mar 28. PMID 12658421
- [Background] Oelschlager BK, Pellegrini CA, Hunter JG, Brunt ML, Soper NJ, Sheppard BC, Polissar NL, Neradilek MB, Mitsumori LM, Rohrmann CA, Swanstrom LL. Biologic prosthesis to prevent recurrence after laparoscopic paraesophageal hernia repair: long-term follow-up from a multicenter, prospective, randomized trial. J Am Coll Surg. 2011 Oct;213(4):461-8. doi: 10.1016/j.jamcollsurg.2011.05.017. Epub 2011 Jun 29. PMID 21715189
- [Background] Velanovich V. The development of the GERD-HRQL symptom severity instrument. Dis Esophagus. 2007;20(2):130-4. doi: 10.1111/j.1442-2050.2007.00658.x. PMID 17439596
- [Derived] Petro CC, Ellis RC, Maskal SM, Zolin SJ, Tu C, Costanzo A, Beffa LRA, Krpata DM, Alaedeen D, Prabhu AS, Miller BT, Baier KF, Fathalizadeh A, Rodriguez J, Rosen MJ. Anterior Gastropexy for Paraesophageal Hernia Repair: A Randomized Clinical Trial. JAMA Surg. 2025 Mar 1;160(3):247-255. doi: 10.1001/jamasurg.2024.5788. PMID 39714889
- [Derived] Blake KE, Zolin SJ, Tu C, Baier KF, Beffa LR, Alaedeen D, Krpata DM, Prabhu AS, Rosen MJ, Petro CC. Comparing anterior gastropexy to no anterior gastropexy for paraesophageal hernia repair: a study protocol for a randomized control trial. Trials. 2022 Jul 30;23(1):616. doi: 10.1186/s13063-022-06571-8. PMID 35907909